CLINICAL TRIAL: NCT03950479
Title: Pelvic Floor Muscle Assessment at 3-and 4-dimensional Transperineal Ultrasound and Its Relation to Pregnancy and Labor
Brief Title: Pelvic Floor Muscle Assessment at 3-and 4-dimensional Transperineal Ultrasound
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, Assistant professor of obstetrics and gynecology, Cairo University
Other Study IDs: pelvic floor
Record Dates: First submitted 2019-05-11; First posted 2019-05-15 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- primiparous group: women who will give birth to their first baby
  Interventions: Diagnostic Test: 3D and 4D Transperineal Ultrasound

INTERVENTIONS:
Diagnostic Test: 3D and 4D Transperineal Ultrasound — The evaluation of Pelvic Floor Muscles with 3D and 4D transperineal ultrasound using A Voluson E6 system (GE Healthcare, Zipf, Austria) with RAB 8-4-MHz volume transducer for all acquisitions. Measurements will be performed in axial planes. The levator hiatus area (LHA), the antero-posterior (AP) diameter and the left-right (LR) transverse diameter will be analyzed at rest, during pelvic floor contraction and on maximal Valsalva maneuver.

SUMMARY:
Injuries to the pelvic floor muscles and fascias during delivery and childbirth may lead to urinary incontinence (25-45 %), faecal incontinence (11-45%), pelvic organ prolapse (7-23%), sexual dysfunction (15-33 %) and chronic pain syndromes (4-15%). Pelvic floor muscle injuries are not easy to diagnose as they are not visible when looking at surface anatomy during a standard gynaecological examination. The investigators are therefore in urgent need of better tools to diagnose these injuries. Having a reliable and easily accessible tool enables studies of the consequences of such pelvic floor muscle injuries. It also makes it possible for us to explore the effect of interventions such as pelvic floor muscle training and surgery in patients with and without pelvic floor muscle injuries. The investigators have previously presented data to support the reliability and the validity of the three and four dimensional (3 and 4D) ultrasound technique used to define pelvic floor muscle anatomy in healthy volunteers and have now a tool to study women before and after delivery.

DETAILED DESCRIPTION:
At the Department of Obstetrics and Gynaecology, Cairo University Hospital there are approximately 29000 deliveries annually and 10000 women are giving birth for the first time.

Challenges: The invitation to participate in the study will be given to all women expecting their first child fulfilling inclusion criteria. The biggest challenges in the project will be logistical. To be able to inform, recruit and follow women having their first child is a challenge in itself.

Applications: If it is possible to identify a risk group for pelvic floor injuries before delivery, it might be ethical to recommend a prophylactic cesarean section to avoid disabling incontinence and prolapse later in life.

ELIGIBILITY:
Inclusion Criteria:

* Women giving birth to their first child at Cairo University Hospital, Egypt and University Hospital Würzburg, Germany.

Exclusion Criteria:

* Previous pregnancy of more than 16 weeks.
* preterm delivery less than 32 weeks gestation.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women giving birth to their first child at Cairo University Hospital, Egypt and University Hospital Würzburg, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Levator Hiatus Area at Rest Measured Via 3-dimensional transperineal Ultrasound at Gestational Week 24 and 37 | 24 weeks and 37 weeks of gestation
  3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Levator hiatus area was measured at gestational week 24 and 37, at rest, during contraction and during Valsalva maneuver - giving 6 measurements all together. The change in LH area was computed between the two different timepoints giving 3 outcomes

SECONDARY OUTCOMES:
Change in Levator Hiatus Area at Contraction Measured Via 3D transperineal Ultrasound at Gestational Week 24 and 37 | 24 weeks and 37 weeks of gestation
  3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Levator hiatus area was measured at gestational week 24 and 37, at rest, during contraction and during Valsalva maneuver - giving 6 measurements all together. The change in LH area was computed between the two different timepoints.
Change in Levator Hiatus Area During Valsalva Maneuver Measured Via 3D transperineal Ultrasound | gestational week 24 and 37
  3-dimensional ultrasound was used to capture the axial plane of the pelvic floor in order to measure LH area. Levator hiatus area was measured at gestational week 24 and 37, at rest, during contraction and during Valsalva maneuver - giving 6 measurements altogether. The change in LH area was computed between the two different timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — Cairo University